CLINICAL TRIAL: NCT05335512
Title: Intravesical BCG: is the Urinary Bladder Ready to Receive it
Status: Not yet recruiting | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr. Mahendra Pal, Professor Urology Oncology, Tata Memorial Centre
Other Study IDs: 3505
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Non-Invasive Bladder Urothelial Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent TURBT: Patients undergoing complete TURBT for evaluation of a newly diagnosed bladder lesion in TMH and found to have NMIBC (either low risk or high risk)

SUMMARY:
Prospective cohort and Prospective observational study which aims To define the healing time-frame of the resected area of the bladder after TURBT. and also to validate a grading system of healing of the bladder mucosa after TURBT. To assess the factors influencing bladder healing is also one of the secondary objectives.

DETAILED DESCRIPTION:
This study will be offered to patients who are coming to Tata Memorial Hospital (TMH) for management of Non Muscular Invasive bladder cancer. 10 patients who undergo Transurethral resection of Bladder tumour will be enrolled. Any patient who undergoes TURBT in TMH, found to have NMIBC and gives consent is eligible for the study. Patient who has visible tumor on first or any subsequent cystoscopy are not eligible.

100 patients (40 private category & 60 general category patients) will be recruited, and they will be planned for cystoscopy in the minor operation theater under antibiotic cover and local anaesthesia at 2nd week, 3rd week, 4th week after the date of TURBT.

Apprehensive or uncooperative patient will undergo procedure under general anaesthesia.

Patients having non healed bladder mucosa at 4 weeks will be reassessed after a further 1week by additional cystoscopy.Each time of cystoscopy a photo of the healing resected area will be captured and will be used to compare with the next photo in the same patient to see the progress of healing. These photos will be assess by two experienced uro-oncologist to characterize the healing status of bladder.This comparison will be used to establish a grading system of bladder healing. The remaining cystoscopies will be performed as per guidelines. Urine routine microscopy and culture/sensitivity will be done before every cystoscopy to rule out urinary tract infection and to quantify the numbers of white blood cells the WBC count will be correlated with the degree of inflammation and phases of healing as additional marker. Patients who have healed or near healed resection area on any cystoscopy as per study protocol will be given IVB in the same setting if the patient is stratified as high risk NMIBC. Patients who will be stratified as low-risk NMIBC and has healed resection area will not have further cystoscopy as per study protocol but will undergo cystoscopy later as per guideline's schedule. Any patient having unhealed resection on cystoscopy will be planned for next cystoscopy as per protocol and IVB will not be given at this cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing complete TURBT for evaluation of a newly diagnosed bladder lesion in TMH and found to have NMIBC (either low risk or high risk) Patient gives consent will be included (after explaining about the study).

Exclusion Criteria:

1. Patient who has visible tumor on first or any subsequent cystoscopy.
2. On histopathology found to have muscle invasive bladder cancer.
3. Patient having urinary tract infection before cystoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be offered to patients who are coming to Tata Memorial Hospital (TMH) for management of NMIBC.
  Approx 10 patients who undergo TURBT in TMH will be enrolled in the pilot study as per study design. Based on validation of result of this study, proposed study will be carried out that will have 100 patients with same method including 10 patients of pilot study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Time Frame after TURBT | 1 year
  To define the healing time-frame of the resected area of the bladder after TURBT.

SECONDARY OUTCOMES:
Validate Grading System | 1 year
  The score is from grade 1 to grade 4, the title for grading 'Grading of healing with time', minimum value 1 is while maximum value 4 is and higher scores means a worst outcome
Assessment Factors | 1 year
  To assess the factors influencing bladder healing.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers but overall data will be published after the study completion.